CLINICAL TRIAL: NCT07037992
Title: The Effect of Subcostal Anterior Quadratus Lumborum Block on the Incidence of Chronic Neuropathic Pain After Retroperitoneal Laparoscopic Donor Nephrectomy: A Study on Neuroinflammation and Neurophysiology
Brief Title: The Effect of Quadratus Lumborum (QL) Block on the Incidence of Chronic Neuropathic Pain After Retroperitoneal Laparoscopic Donor Nephrectomy: A Study on Neuroinflammation and Neurophysiology
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Raden Besthadi Sukmono, Anesthesiologist, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLChronicNeuropathicPostOpPain
Record Dates: First submitted 2025-05-26; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Living Kidney Donor; Quadratus Lumborum Block; Laparoscopic Donor Nephrectomy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (Experimental)
  Interventions: Drug: injection of local anesthesia solution
- Quadratus Lumborum Sham Block (Placebo Comparator)
  Interventions: Drug: Injection of normal saline

INTERVENTIONS:
Drug: injection of local anesthesia solution — Injection of 30 mL local anesthetic solution bupivacaine 0.25%
  Arms: Quadratus Lumborum Block
Drug: Injection of normal saline — Injection of 30 mL normal saline Natrium Chloride (NaCl) 0.9%
  Arms: Quadratus Lumborum Sham Block

SUMMARY:
To analyze the relationship of anterior subcostal quadratus lumborum (QL) block compared with control block on the incidence of chronic neuropathic pain at three months post-laparoscopic retroperitoneal living kidney donor.

ELIGIBILITY:
Inclusion Criteria:

Living kidney donor candidate patients aged 18-65 years Patients with ASA physical status assessment 1-3 Patients are willing to be research subjects.

Exclusion Criteria:

* The patient was known to have a history of chronic non-cancer pain and cancer pain.

The patient had a history of preoperative laparoscopic kidney donor surgery.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Neuropathic Pain Incidence: Neuropathic Pain in 4 Questionnaire | 3 months after intervention
  Pain that develops after a surgical procedure in the area of surgery and its radiation, persists for at least 3 months after surgery, other causes of pain (e.g. infection and history of malignancy) or pre-existing pain have been excluded.
  Total score: 10 Score ≤ 4 = no pain developed Score ≥ 4 = pain developed
Neuromodulation Parameter: Degree of functional interference using Behavioral Pain Interference (BPI) | At 3 months after intervention
  The degree of pain that develops after a surgical procedure in the area of surgery and its radiation, persisting for at least 3 months after surgery, other causes of pain (eg infection and history of malignancy) or pre-existing pain have been excluded.
  Behavioral Pain Interference (BPI) questionnaire based on the average of questions 4, 5, and 6
  1. Mild (NRS 1-3)
  2. Moderate (NRS 4-6)
  3. Severe (NRS 7-10)
Chronic Pain Severity: Leeds Assesment of neuropathic symptoms and sign (LANSS) scale | At 3 months after intervention
  A measuring tool used to assess neuropathic pain and provides information to differentiate nociceptive pain from neuropathic pain.
  Total score: 24 <12: Not neuropathic >12: Neuropathic pain
Neuroinflammation Parameter: Serum Concentration of Toll-like Receptor 4 (TLR4) | At 3 months after intervention
  Transmembrane receptors in the innate immune system. Units: ng/mL
Neuroinflammation Parameter: Serum Concentration of Calcitonin gene-related peptide (CGRP) | At 3 months after intervention
  Neuropeptides that play a role in pain transmission and vasodilation Unit: pg/mL
Neuroinflammation Parameter: Serum Concentration of Nerve Growth Factor (NGF) | At 3 months after intervention
  Neurotrophic factors that play a role in promoting the growth and survival of sensory neurons Unit: pg/mL
Neurophysiology Parameter: Mechanical Detection Threshold (MDt) | At 3 months after intervention
  Measures the minimum force needed for a person to perceive a light mechanical stimulus, tested using von Frey filaments. Skin contact test for 2 seconds using 1 set of von Frey filaments. The examination is performed in m. trapezius.
  Unit: mN Lower result means: higher sensitivity (normal or hypersensitivity) Higher result means: Reduced sensitivity, could indicate hypoesthesia or nerve damage
Neurophysiology: Mechanical Pain Threshold (MPt) | At 3 months after intervention
  Accurate measurement of pain threshold. Skin contact test using repeated pinpricks at the same location. Comparative assessment of initial pain scale with pain scale after repeated stimulation. Examination is performed at m. trapezius.
  Unit: Numerical Rating Scale (NRS) from 1 to 10 Lower NRS: higher sensitivity to pain Higher NRS: lower sensitivity to pain
Neurophysiology Parameter: Pressure Pain Threshold (PPt) | At 3 months after intervention
  Pain tolerance examination. Pressure assessment in kgf/cm2 units where the patient complains of pain according to the stimulus given. The examination is carried out in m. trapezius Units: kgf/cm2.
  Lower PPT: Increased pain sensitivity Higher PPT: Decreased pain sensitivity
Neurophysiology Parameter: Mechanical Temporal Summation of Pain (MTSP) | At 3 months after intervention
  Evaluates central sensitization by applying repeated light mechanical stimuli and rating how pain builds up over time.
  Pressure assessment in kgf/cm2 units where the patient complains of pain according to the stimulus given. The examination is carried out in m. trapezius.
  Units: Verbal Numeric Scale (VNS) from 1 to 10 Higher MTSP score: Indicates central sensitization Lower MTSP score: Normal pain processing
Neuromodulation Parameter: Serum Concentration of beta-Endorfin | At 3 months after intervention
  Neuropeptide produced in the anterior pituitary and brain, as an endogenous opioid.
  Units: pg/mL

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No